CLINICAL TRIAL: NCT03614754
Title: The Involvement of Pudendal Somatic Afferents in Sacral Neuromodulation Assessed by Somatosensory Evoked Potentials of the Pudendal Nerve
Brief Title: Sacral Neuromodulation and Pudendal Somatic Afferents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Donald Vaganée, MD, PhD student, Universiteit Antwerpen
Other Study IDs: 17/30/334
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Overactive Bladder, Non Obstructive Urinary Retention
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Evoked Potentials, Somatosensory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successes: Patients with reduction of symptoms >50% during the test procedure for sacral neuromodulation.
  Interventions: Diagnostic Test: Somatosensory evoked potentials
- Failures: Patients with reduction of symptoms <50% during the test procedure for sacral neuromodulation.
  Interventions: Diagnostic Test: Somatosensory evoked potentials

INTERVENTIONS:
Diagnostic Test: Somatosensory evoked potentials — Stimulation of the pudendal nerve while recording at the sensory cortex.

SUMMARY:
Sacral neuromodulation is a well-excepted minimally invasive procedure for the treatment of overactive bladder and non-obstructive urinary retention.A tined lead with 4 stimulation electrodes is placed through the third or fourth sacral foramen and stimulates sacral roots in its vicinity. Since the sacral roots are mixed nerves, it is currently still unknown which nerve fibers are stimulated (autonomic vs somatic, afferent vs efferent) and what the mechanism of action is.

This study examines the involvement of pudendal somatic afferents by measuring somatosensory evoked potentials elicited by stimulation of the pudendal nerve.

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder
* Non-obstructive urinary retention

Exclusion Criteria:

* Neurogenic disorders (e.g. cerebrovascular accident, spinal cord injury,...)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Urological patients with overactive bladder or non-obstructive urinary retention.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Latency change | 3 weeks
  Latency of somatosensory evoked potential are recorded before and after test procedure sacral neuromodulation expressed in milliseconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided